CLINICAL TRIAL: NCT00963001
Title: Effect of Different Meal Types on the Pharmacokinetics of a Single 1 mg Oral Dose of UT-15C (Treprostinil Diethanolamine) Sustained Release Tablets in Healthy Volunteers
Brief Title: Effect of Food on the Pharmacokinetics of Oral Treprostinil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Allison Pecha, United Therapeutics Corp.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-115
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Hypertension, Pulmonary; Pulmonary Arterial Hypertension
Keywords: Hypertension, Pulmonary; Treprostinil; Pharmacokinetics; Treprostinil Diethanolamine; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Treprostinil diethanolamine — Subjects will each receive a single 1 mg sustained release tablet of treprostinil diethanolamine by mouth within 10 minutes of consuming each of four standardized meals on Study Days 1, 8, 15, and 22.
  Other Names: UT-15C; UT-15C SR; Oral treprostinil
Other: Standardized meals — Each subject will receive one of four different standardized meals of varying caloric and fat content in a randomized sequence such that all subjects will receive all four meals over the course of the study. Each subject will receive one standardized meal for breakfast on Study Days 1, 8, 15, and 22.

SUMMARY:
The purpose of this study is to assess the pharmacokinetic and safety profile of a single dose of oral treprostinil following four different meals of varying caloric and fat content.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy and between the ages of 18 and 55 years, inclusive, at Screening.
* Female subjects must weigh between 45 and 100 kg, inclusive, with a BMI between 19.0-29.9 kg/m2, inclusive at Screening. Male subjects must weigh between 50 and 120 kg, inclusive, with a BMI between 19.0-32.0 kg/m2, inclusive at Screening.
* Subject has a medical history, physical examination, vital signs, ECG and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at Screening.

Exclusion Criteria:

* Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations.
* Subject has a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
* Subject has a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Treprostinil pharmacokinetics in healthy volunteers following a single oral dose of a 1 mg treprostinil diethanolamine sustained release tablet after four different meal types. | Immediately prior to through 36 hours post treprostinil diethanolamine dosing for each treatment period (4 treatment periods each separated by a 7-day washout period)
Adverse event monitoring | From the first dose of treprostinil diethanolamine through study end (Study Day 23/24)

SECONDARY OUTCOMES:
Clinical laboratories | Study Days 0, 7, 14, 21 and 23

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Laurent, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, Austin, Texas, United States